CLINICAL TRIAL: NCT07373470
Title: Genotype-guided Comprehensive Medication Management to Improve Depression Outcomes in Pennsylvania
Brief Title: An Evaluation of the Impact of Pharmacist Comprehensive Medication Management With Pharmacogenomic Results to Improve Depression Outcomes in Community Pharmacies.
Acronym: COMPASS-PGx
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Pennsylvania Department of Health (Other Government)
Responsible Party: Principal Investigator, Philip Empey, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY21120100
Record Dates: First submitted 2026-01-12; First posted 2026-01-28 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Pharmacogenetics; Depression - Major Depressive Disorder; Pharmacogenomic Drug Interaction; Community Pharmacy Services
Keywords: precision medicine; pharmacogenomics; PGx; Comprehensive medication management; pharmacist; community pharmacy; medication review; antidepressants; pharmacogenomic testing; management of depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive medication management with PGx testing results (Experimental): Participants will have a study visit with a community pharmacist for comprehensive medication management with review of PGx testing results.
  Interventions: Other: Comprehensive medication management with PGx testing results
- Usual care (Other): Participants will receive no study intervention (usual care) and will have a comprehensive medication management with review of PGx testing results at the end of the study.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Comprehensive medication management with PGx testing results — A comprehensive medication management with PGx testing includes a pharmacist-provided review of health history, past/current medications, and assessment of potential medication related problems. A review of PGx testing results will be integrated to identify any PGx-related medication issues. Recommendations will then be made to study participants' providers (regular care team) for any decisions regarding potential therapy changes.
  Arms: Comprehensive medication management with PGx testing results
Other: Usual Care — Participants will receive no study intervention (usual care) and will have a comprehensive medication management with review of PGx testing results at the end of the study.
  Arms: Usual care

SUMMARY:
The goal of this prospective, randomized clinical trial is to learn whether pharmacogenomic (PGx)-guided comprehensive medication management delivered by pharmacists in community pharmacies will improve antidepressant treatment outcomes.

The primary aim is to determine whether comprehensive medication management with review of PGx testing results improves depression symptoms, compared with usual care.

Participants 18 years of age or older who have undergone PGx testing (e.g. through an independent biobanking study (Pitt+Me Discovery) who require initiation or adjustment of antidepressant therapy will be randomly assigned to receive either PGx-guided comprehensive medication management or usual care. Those who receive usual care will receive their PGx results at the end of the study. Researchers will compare the groups to assess whether PGx-guided care provided in partnership with community pharmacists and prescribers results in better depression and medication outcomes.

ELIGIBILITY:
INCLUSION CRITERIA:

* At targeted community pharmacy for:

  * New prescription or change in dose/schedule of SSRI (citalopram, escitalopram, sertraline, paroxetine), OR
  * Concurrent SSRI (citalopram, escitalopram, sertraline, paroxetine) and new prescription/change in SNRI (desvenlafaxine, duloxetine, and venlafaxine) / bupropion.
* Depressive symptoms confirmed by PHQ8 assessment (>5 indicating at least mild depressive symptoms)
* UPMC patient (or able/willing to become one) and has UPMC provider (or able/willing to obtain one)
* Signed consent to join Pitt+Me Discovery biobanking research study.
* English-speaking

EXCLUSION CRITERIA:

* Inability to receive CMM at specific pharmacy/pharmacist
* Comorbid diagnosis of schizophrenia (patient-reported)
* Untreated sleep disorder (patient-reported)
* Pitt+Me Discovery participant who has elected to not receive return of results, or who has already received results previously

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire (PHQ-8) score | Baseline, 6 Weeks, 12 Weeks, 6 Months
  The Patient Health Questionnaire-8 (PHQ-8) is an 8-item self-report measure assessing depressive symptoms. Each item is scored from 0-3, producing a total score of 0-24, with higher scores indicating more severe depressive symptoms. Standard severity categories are minimal (0-4), mild (5-9), moderate (10-14), moderately severe (15-19), and severe (20-24).

SECONDARY OUTCOMES:
Change in the Extent of Adherence and Reasons for Nonadherence Survey (Voils et al.) score | Baseline, 6 Months
  The Extent of Adherence and Reasons for Nonadherence Survey (Voils et al.) is a validated self-report measure assessing medication adherence over the past 7 days. It is scored on a 1-5 Likert scale and averaged to produce a continuous score, with higher scores indicating better adherence. The Reasons for Nonadherence scale assesses specific barriers to taking medication as prescribed, with items rated on a 1-5 scale and assessed individually to identify the degree to which each barrier contributed to missed doses.
Change in Generalized Anxiety Disorder Assessment (GAD-7) score | Baseline, 6 Weeks, 12 Weeks, 6 Months
  The Generalized Anxiety Disorder Assessment (GAD-7) is a 7-item self-report measure assessing anxiety symptoms over the past two weeks, with items scored 0-3 for a total score of 0-21; higher scores indicate more severe anxiety, categorized as minimal (0-4), mild (5-9), moderate (10-14), and severe (15-21).
Proportion of pharmacist recommendations were accepted | 6 months
  Proportion of pharmacist recommendations to address medication-related problems that were accepted by providers as assessed by EHR and fill data review.
Change in frequency of CPIC/FDA guideline concordant prescribing | Baseline, 6 Months
  Change in frequency of concordance of participant medication regimen with pharmacogenomics prescribing recommendations according to the Clinical Pharmacogenomics Implementation Consortium (CPIC) and U.S. Food & Drug Administration (FDA) guidelines using electronic health record data.
Number of adverse events as assessed using the Frequency, Intensity, and Burden of Side Effect rating scale (FIBSER). | Baseline, 6 Weeks, 12 Weeks, 6 Months
  The Frequency, Intensity, and Burden of Side Effect Rating Scale (FIBSER) is a 3-item self-report measure assessing medication side effects. It evaluates the frequency, intensity, and functional burden of side effects over the past week, with each item rated on a 0-6 scale; higher scores indicate more frequent, severe, or burdensome side effects. Clinically, a total score of 0-2 typically requires no change in treatment, 3-4 side effects may warrant targeted management, and 5-6 indicates that treatment modification should be considered to improve tolerability and adherence.
Frequency of Actionable Genotypes | 6 months
  Frequency of actionable genotypes (in the entire study population) based on report of a genotype-predicted phenotype. Actionable genotypes are defined as those with recommendations for a change in prescribing by a CPIC (Clinical Pharmacogenetics Implementation Consortium) guidelines or FDA recommendations.
Number of participant medications with PGx guidance based on PGx testing results. | 6 months
  This measure counts the number of a participant's medications for which pharmacogenomic (PGx) guidance is available based on PGx testing results. Medications with PGx guidance may have dosing recommendations, alternative drug options, or monitoring considerations informed by the participant's genetic profile.
Change in healthcare utilization | From Baseline to 6 Months
  Change in participant ER visits, hospitalizations, urgent care visits, specialist appointments, primary care appointments, and unplanned care using UPMC EHR data.

OTHER OUTCOMES:
Community pharmacists' needs for expert support in deploying PGx | 6 Months
  Community pharmacists' needs for expert support in deploying PGx Number and types of questions asked by community pharmacists to PGx experts on study team through the duration of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Philip E Empey, PharmD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No